CLINICAL TRIAL: NCT04432727
Title: A Feasibility Study Evaluating the Impact Flexitouch Plus With Connectivity Has on Compliance in Patients With Breast Cancer-Related Lymphedema (BCRL)
Brief Title: Study Evaluating Flexitouch Plus With Connectivity on Compliance in 30 Patients With Breast Cancer-Related Lymphedema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4090
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ACTIVE FT-CC (Experimental): Text message reminders will be sent if subject does not use the device for 2 consecutive days.
  Interventions: Device: Flexitouch Plus with Cellular Connectivity (FT-CC)
- PASSIVE FT-CC (Experimental): Text message reminders will not be sent to subjects.
  Interventions: Device: Flexitouch Plus with Cellular Connectivity (FT-CC)

INTERVENTIONS:
Device: Flexitouch Plus with Cellular Connectivity (FT-CC) — Daily use of FT-CC

SUMMARY:
The objective of this study is to demonstrate the feasibility of using the Flexitouch Plus with Cellular Connectivity (FT-CC) to monitor device use data to determine if reminders to patients impact compliance, and to identify the impact device compliance has on arm girth, quality of life (QOL), and symptom assessment.

DETAILED DESCRIPTION:
This is a multi-center, on label, prospective, randomized, two-arm feasibility study that plans to enroll 30 female subjects in the United States. In an effort to reduce potential exposure to COVID-19, all study assessments are intended to be performed in a contactless manner (i.e., telephone, video conference, etc). If a subject passes the initial screening requirements via medical history and expresses interest in the study an informed consent form will be provided to them. Once consent has been obtained they will undergo a baseline visit where they will be randomized to one of two treatment groups: PASSIVE FT-CC (text messages reminders will not be sent to subjects) and ACTIVE FT-CC (text messages reminders will be sent if subject does not use the device for 2 consecutive days). Randomization was incorporated into the study to determine if ACTIVE FT-CC affects device use. A total of 2 follow-up visits will be conducted over a 60-day period.

ELIGIBILITY:
Inclusion Criteria:

1. Female 18 years of age or older
2. Diagnosis of unilateral breast cancer-related lymphedema
3. Willing and able to give informed consent (remotely or in person)
4. Willing and able to comply with the study protocol requirements and all study-related visit requirements, including the ability to participate remotely
5. Willing and able to receive text messages from sponsor

Exclusion Criteria:

1. In-home use of PCD within previous 3 months
2. Phase-one CDT within previous 1 month or planned phase-one CDT during study participation Phase-one CDT defined as professionally administered MLD and/or multi-layer short stretch compressive bandaging.
3. Inability to be fit for PCD garments
4. Heart failure (acute pulmonary edema, decompensated acute heart failure)
5. Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)
6. Active skin or limb infection/inflammatory disease (acute cellulitis, other uncontrolled skin or untreated inflammatory skin disease) on the arms or trunk
7. Currently receiving treatment for cancer with curative intent.
8. Any circumstance where increased lymphatic or venous return is undesirable
9. Currently pregnant or trying to become pregnant
10. Known inability to receive cell phone connection where FT-CC therapy will be administered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pesek, MD, Principal Investigator — St. Peter's Health Partners; Nicolas Ajkay, MD, Principal Investigator — University of Louisville
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - St. Peter's Hospital, Albany, New York
  - Samaritan Hospital Hildegard Medicus Cancer Center, Troy, New York

REFERENCES:
- [Derived] Maingi S, O'Malley EM. Impact of text reminders on pneumatic compression device (PCD) compliance in patients with breast cancer-related lymphedema. Support Care Cancer. 2023 Dec 16;32(1):33. doi: 10.1007/s00520-023-08246-9. PMID 38102530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACTIVE FT-CC | PASSIVE FT-CC
Started | 15 | 14
Completed | 14 | 11
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACTIVE FT-CC | PASSIVE FT-CC | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.8) | 57.7 (9.7) | 54.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 15 | 11 | 26
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 13 | 10 | 23
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29
Weight [Mean (Standard Deviation); unit: pounds] | 190.9 (42.8) | 179.1 (42.0) | 185.2 (42.1)
Height [Mean (Standard Deviation); unit: inches] | 63.8 (2.3) | 62.4 (1.6) | 63.1 (2.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.1 (8.0) | 32.4 (7.4) | 32.8 (7.6)
Dominant Hand [Count of Participants; unit: Participants]
  Left | 1 | 1 | 2
  Right | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Compliance Measured as the Average Number of Treatments Per Week
Description: Compare the rate of compliance in patients treated with PASSIVE FT-CC and ACTIVE FT-CC.
Time Frame: 60 Days
Population: Patients who received text reminders vs. those that did not.
Measure: Mean (Standard Deviation); unit: treatments/week
Arm/Group | ACTIVE FT-CC | PASSIVE FT-CC
Number analyzed (Participants) | 15 | 14
treatments/week | 5.3 (1.8) | 5.2 (2.1)

2. Secondary Outcome: Compliance With Device Use.
Description: Analysis of compliance with prescribed device use.
Time Frame: Through 60 days after device training
Population: Subjects who were also seen 60 days post randomization.
Measure: Count of Participants; unit: Participants
Groups:
- ACTIVE FT-CC: Text message reminders were sent if the subject did not use the device for 2 consecutive days. Flexitouch Plus with Cellular Connectivity (FT-CC): Daily use of FT-CC
- PASSIVE FT-CC: Text message reminders were not sent to subjects. Flexitouch Plus with Cellular Connectivity (FT-CC): Daily use of FT-CC
Arm/Group | ACTIVE FT-CC | PASSIVE FT-CC
Number analyzed (Participants) | 13 | 10
Participants
  Non-Compliant (<1 Day / Week) | 0 | 1
  Partially Compliant (1-4 Days / Week) | 6 | 4
  Compliant (5-7 Days / Week) | 7 | 5

3. Secondary Outcome: Quality of Life Assessment Via LYMQOL ARM
Description: Comparison of quality of life in patients treated with Active FT-CC vs. Passive FT-CC via Lymphedema Quality of Life Tool (LYMQOL ARM).
  Lymphedema Quality of Life Tool (LYMQOL-ARM) includes sub-scores for Function (range 10-40), Appearance (range 5-20), Symptoms (range 6-24), and Emotion (range 6-24) where lower scores represent a better outcome. It also includes an Overall QOL sub-score (range 0-10) where a higher score represents a better outcome.
Time Frame: Changes through 60 days after device training
Population: Subjects completing the LYMQOL-ARM Tool at 60 days overall quality of life score 0-10 scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active FT-CC: Subjects receiving text message reminders when device has not been used for 2 days.
- Passive FT-CC: Subjects did not receive text reminders when device was not used.
Arm/Group | Active FT-CC | Passive FT-CC
Number analyzed (Participants) | 14 | 11
score on a scale | 7.6 (2.0) | 6.6 (1.7)

4. Secondary Outcome: Quality of Life Assessment Via SF-36 Physical Functioning Domain Score
Description: Comparison of baseline vs. 60-day follow-up results of the The RAND 36-Item Short Form Survey (SF-36).
  The RAND 36-Item Short Form Survey (SF-36) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item for perceived change in health. Min value: 0, Max value: 100. Higher scores represent a better outcome.
Time Frame: Changes through 60 days after device training
Population: Patients with data through 60 days after device training. An increase in score reflects a positive outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Active FT-CC | Passive FT-CC
Number analyzed (Participants) | 14 | 11
Participants
  Decrease in general health domain scores at 60 days | 4 | 8
  No change in general health domain scores at 60 days | 4 | 0
  Increase in general health domain score change at 60 days | 6 | 3

5. Secondary Outcome: Quality of Life Assessment Via LSIDS-A Score
Description: Comparison of baseline vs. 60-day follow-up results of the LSIDS-A Scoring Tool.
  The LSIDS-A domains consist of 30 questions in the areas of soft tissue sensation, neurological sensation, function, behavior, resource, sexuality, and activity. Scores are compiled by domain and overall. Overall results will be posted here.
Time Frame: Changes through 60 days after device training
Population: All patients with follow-up through 60 days completing the LSIDS-A Questionnaire. A reduction in overall domain score change is considered to be positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Active FT-CC | Passive FT-CC
Number analyzed (Participants) | 13 | 11
Participants
  Decrease in domain score change at 60 days | 12 | 8
  No change in domain score at 60 days | 0 | 0
  Increase in domain score change at 60 days. | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the point of randomization through study exit (Day 60).
Arm/Group | ACTIVE FT-CC | PASSIVE FT-CC
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 4/15 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTIVE FT-CC (N=15) | PASSIVE FT-CC (N=14)
Acute pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTIVE FT-CC (N=15) | PASSIVE FT-CC (N=14)
Clicking in right thumb joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exacerbation of lymphedema related pain right arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suspected cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Trauma secondary to fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphedema exacerbation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Progressive disease right axilla (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Swelling under right arm due to weight gain, no lymphedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Increased lung nodule from 2011 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tender in armpit when using device (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Worsening lymphedema (mild) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic resulted in the closure of several clinics and when clinics were able to resume operations, it was on a limited basis to keep patients and providers physically distanced from others. In addition, reduction of staff impacted research conduct. Finally, patients were often not willing to attend study visits. These factors all contributed to slow enrollment and a high early withdrawal rate which led to the decision to discontinue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT04432727/Prot_SAP_000.pdf